CLINICAL TRIAL: NCT06958471
Title: The Effect of Individualized Developmental Care Education Given to Mothers of Premature Infants on Maternal Self-Efficacy and Attachment Levels
Brief Title: The Effect of Individualized Developmental Care Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Emel AVÇİN, Lecturer Dr, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Emel Avcin Indı. Deve. Care
Record Dates: First submitted 2025-04-18; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Premature; Self Efficacy; Attachment; Maternal
Keywords: Premature; Individualized Developmental Care; Attachment; Self Efficacy; Maternal
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Randomized controlled and Quasi-experimental research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Developmental Care Education Group (Experimental): Before the mother is discharged from the hospital after delivery (within 24 hours for a vaginal birth and within 72 hours for a cesarean section), a brochure titled "Your Premature Baby" prepared by the researcher will be provided. The content of the "Infant Care and Nutrition" booklet to be given to mothers will include information on breastfeeding, infant care, home environment, screening tests, immunization, common problems, and other related topics.
  In the second and third weeks, individualized developmental care training tailored to the needs of the newborn will be provided. This training will cover topics such as environmental adjustments (light, noise, temperature), kangaroo care, infant massage, non-nutritive sucking, and parent-infant bonding.
  In the fourth week, the mothers' application of the training and their knowledge levels regarding premature infant care will be assessed.
  Interventions: Behavioral: Individualized Developmental Care Education Group
- Control group (No Intervention): During the hospitalization of the premature infant, routine nursing education provided in the clinic will be delivered to the mother by the unit nurse. These routine trainings and information sessions include the following:
  A brief information session of approximately 5 minutes, usually given to all mothers within the first 24 hours after birth, covering topics such as breast milk expression, breastfeeding positions, and the benefits of breast milk. Mothers selected for kangaroo care are given information regarding hand hygiene and personal cleanliness.
  On weekdays, between 1:00 p.m. and 2:00 p.m., the neonatologist provides information to parents about the general condition of their baby in the NICU.
  To prevent ethical concerns arising from the implementation of the study in terms of the control group, after the posttest is completed, the researcher will provide the control group families with the information they need.

INTERVENTIONS:
Behavioral: Individualized Developmental Care Education Group — An educational program will be implemented for the mothers in the intervention group throughout the hospitalization period of their premature infants, in line with the objectives of the study.
  P1:Pretests for the mothers will be completed within the first three days of the infant's admission to the neonatal intensive care unit (NICU). Mothers will be given a brochure titled "Your Premature Baby", prepared by the researcher, which includes information about the NICU and its staff, visiting hours/conditions, and breast milk expression times.
  P2:Education will be provided on the characteristics, feeding, and care of premature infants.
  P3:Mothers will receive training on environmental regulations (temperature, light, sound), kangaroo care,non-nutritive sucking, and parent-infant interaction. Each training session will be delivered each lasting no longer than 30-45 minutes.
  P4:A final training session will be provided on home care for the premature infant.
  Arms: Individualized Developmental Care Education Group

SUMMARY:
This study aims to evaluate the effect of individualized developmental care education provided to mothers of premature infants on maternal self-efficacy and maternal-infant attachment. Premature birth can be a stressful and anxiety-inducing experience for mothers, which may negatively impact their self-confidence and ability to establish an emotional bond with their baby.

Structured and individualized developmental care education provided in the neonatal intensive care unit (NICU) enhances mothers' knowledge and promotes their active participation in the care process, thereby strengthening their maternal roles. Increased self-efficacy helps mothers to take a more active and conscious role in their infant's care, while stronger maternal attachment plays a critical role in the infant's emotional and neurodevelopmental health.

Therefore, the integration and dissemination of such supportive educational interventions within the healthcare system are essential steps that can positively influence both maternal and infant health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The mother must have a premature baby born between 22 and 32 weeks gestation, admitted to a level 3 NICU.
* The baby's stay in the level 3 NICU must be at least one month.
* The mother must not have any diagnosed psychiatric disorders.
* The baby must not have severe congenital anomalies incompatible with life.
* The mother must be literate and open to communication.
* The mother must be willing and volunteer to participate in the research.

Exclusion Criteria:

* The baby's stay in the NICU must be at least one month.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The sample consists of mothers whose premature babies are hospitalized in the NICU.
Enrollment: 60 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Self-Efficacy | The first three days of hospitalization and one month after hospitalization
  Pretests will be administered within the first three days of the mother's admission to the hospital with her premature infant, and posttests will be conducted at the end of the first month. The General Self-Efficacy Scale consists of 17 items. The total score can range from 17 to 85; higher scores indicate a greater belief in self-efficacy.
Maternal Attachment Levels | The first three days of hospitalization and one month after hospitalization
  Pretests will be administered within the first three days of the mother's admission to the hospital with her premature infant, and posttests will be conducted at the end of the first month. The Maternal Attachment Scale consists of 26 items. The total score can range from 26 to 104; higher scores indicate a stronger level of maternal attachment.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL AVÇİN, Doctor, Principal Investigator — University of Yalova
Locations (1):
- Emel Avçin, Yalova, Turkey (Türkiye)